CLINICAL TRIAL: NCT00284245
Title: Internet-based Study of 10,000 Subjects With Chronic Pain, Including Subject-drawn Pain Diagrams, and Computer-generated Composite Images of Pain Patterns
Brief Title: Evaluation of Pain Location, Pain Quality and Pain Patterns in Subjects With Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taylor MicroTechnology (Industry)
Responsible Party: Colin R Taylor, Taylor MicroTechnology, Inc.
Other Study IDs: TMT-B-011; 04076-01; NCT00915395 (obsolete NCT alias)
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2006-09

CONDITIONS: PAIN; CHRONIC DISEASE
Keywords: Chronic Pain; Pain; Computer Analysis; Pain Diagrams
MeSH Terms: conditions — Pain; Chronic Disease; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In earlier work, the Sponsor developed a computer image processing system for analysis of pain diagrams from patients with chronic pain. This system was then tested in a study in over 500 chronic pain patients seen by both primary care practitioners and pain specialists. The hypothesis was that pain location would correlate with the pain type and the underlying cause of the pain. In the study, the computer analysis demonstrated clear correlations between pain diagram data and diagnosis/pain type. The present study extends these observations in a web-based setting, with a focus on the value of computer analysis of pain diagrams as diagnostic predictors.

DETAILED DESCRIPTION:
Earlier work performed by the Sponsor (TMT) included development of a MatLab/ImageJ computer image processing system for generation of composite images from pain diagrams drawn by patients with pain, and for calculation of related quantitative variables. The system was tested in a pharmaceutical company-sponsored US study in over 500 chronic pain patients seen by primary care practitioners, and then seen by pain specialists. The hypothesis was that pain location would correlate with the pain type and the underlying cause of the pain. TMT's analysis established correlations between the pain diagram information and the underlying diagnosis and pain type (e.g., nociceptive or neuropathic) reported by the pain specialists. The present study extends these observations in a web-based setting, with particular emphasis on automated computer-generated visual pain patterns as diagnostic predictors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 18 years of age and of legal age of consent for the state in which they live.
* Able to respond to a questionnaire written in English.
* Report chronic pain (constant or recurring pain lasting more than 30 days and causing significant discomfort or limitation of activity).
* Provide informed consent to participate in the study.

Exclusion Criteria:

* Currently participating in another clinical trial.
* Institutionalized person such as a prisoner or nursing home resident.
* Questionnaire response suggests a medical or psychological condition that, in the opinion of the investigator, would compromise participation in the study, or suggests any other condition which, in the investigator's judgment, might increase the risk to the subject or decrease the chance of obtaining valid data.
* Pain has resulted in a workman's compensation case.
* Pain has resulted in litigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers recruited in Internet study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Colin R Taylor, MD, Principal Investigator — Taylor MicroTechnology, Inc.
Locations (1):
- Taylor MicroTechnology, Inc., New York, New York, United States

REFERENCES:
- See also: Home Page for TMT — http://masterdocs.com
- See also: Background information on study — http://masterdocs.com/chronic_pain_survey__introduction.htm
- See also: Informed Consent Form required before subject enters study — https://www.masterdocs.com/informed_consent_form.htm